CLINICAL TRIAL: NCT06916455
Title: Evaluation of the Nutritional Status of Omega-3 Fatty Acids and the Possible Influences of Dietary Patterns and Different Socioeconomic Factors in a Spanish Population Over 60 Years of Age
Brief Title: Evaluation of the Nutritional Status of Omega-3 Fatty Acids and the Possible Influences of Dietary Patterns and Different Socioeconomic Factors, in a Spanish Population Over 60 Years of Age
Acronym: OMEGAPRED
Status: Recruiting | Type: Observational
Sponsor: Universidad de Granada (Other)
Collaborators: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, María Dolores Mesa García, Proffesor, Universidad de Granada
Other Study IDs: OMEGAPRED (PIP-0265-2024); PIP-0265-2024 (Other: Junta de Andalucía)
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Fatty Acids, Omega-3
Keywords: erythrocyte omega-3 fatty acids; population over 60 years of age; nutritional status; cardiovascular risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, plasma, erythrocytes, white blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Validation cohort: Healthy people (n=200) over 60 year of age that will be bleeded for the validation of the dry spot methodology
- Exploratory cohort: Healthy people (n=600) over 60 year of age that will be study with the dry spot methodology

SUMMARY:
The long-chain polyunsaturated fatty acids (PUFA) of the n-3 or omega-3 series and, in particular, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), both derived from the essential fatty acid alpha-linolenic acid, are part of all cell membranes and from them derive numerous compounds such as prostaglandins, thromboxanes, leukotrienes, resolvins, protectins and maresins that play numerous biological roles, most notably in the control of body homeostasis, blood coagulation and inflammation. The omega-3 index is a biomarker that reflects the nutritional status of n-3 PUFA, as well as cardiometabolic risk and cardiovascular health. This index is determined as the sum of the percentages in weight of EPA and DHA over the total of fatty acids present in the erythrocyte membranes.

Previous studies carried out in Spain, such as ANIBES, indicate that in adults, and especially in those over 60 years of age, the intake of n-3 PUFA is well below the international recommendations, which is directly related to a low intake of fish, since both EPA and DHA are abundant in oily fish. However, in Spain, the nutritional status of omega-3 PUFA and their possible association with a higher prevalence of cardiometabolic risk is unknown, as well as the relationships with food intake and the cultural and socioeconomic status of the population. Therefore, the main objective of the present study is to evaluate the omega-3 index in the Spanish population over 60 years of age and to establish whether there are differences by sex, as well as in the different Spanish communities. In addition, we will study the possible associations between the omega-3 index and food intake, particularly of fish and omega-3 PUFA-rich supplements, as well as their possible associations with cardiometabolic risk indicators and cultural and socioeconomic conditions of the population.

Determination of the omega-3 index usually requires an invasive venous blood collection followed by processing for separation of erythrocytes and extraction and methylation of their membrane lipids followed by chromatographic analysis. But fatty acids can also be determined on whole blood using less invasive methods, such as obtaining drops of blood with a lancet and depositing them on chromatographic paper impregnated with an antioxidant (dried spots). All this makes sampling much easier, although the result of the omega-3 index has to be corrected because it is affected by the lipid composition present in the plasma. For this reason, this project aims to carry out a validation study between the results of the fatty acid profile obtained in erythrocytes and in whole blood in the Spanish population (medamediantedried spots). In short, the results obtained will be used to calculate regression lines that allow us to evaluate the omega-3 index in erythrocytes in the adult Spanish population from different regions of Spain by means of a minimally invasive methodology. For this purpose, 800 participants aged 60 years or more will be recruited from different regions of Spain, randomized by age and sex for each region; at least 100 of the total number of participants should be frequent consumers of omega-3 supplements; if this figure is not obtained, an active search will be carried out until this number is reached (booster). All of them will be interviewed to complete different questionnaires on cultural and socioeconomic status, history of metabolic disease and cardiovascular health, and questionnaires on frequency of consumption and food intake reminders as established by the European Union. With the help of health personnel from different pharmacies and in mutual agreement with the General Council of Pharmaceutical Associations of Spain, a whole blood sample will be taken by lancet, which will be used to quantify the omega-3 index. For the validation study it will be necessary to obtain whole venous blood extracted by venipuncture from a subsample of 200 participants. This sample will be processed and will be used to determine the fatty acid profile in whole blood and in erythrocytes, which will be related by means of multiple linear and bivariate regression models with the fatty acid profile obtained in the dried spots. Cardiometabolic risk markers will also be determined in these 200 subjects, which will be used to establish relationships with the calculated omega-3 status.

ELIGIBILITY:
Inclusion Criteria:

* Older than 60 years of age

Exclusion Criteria: Diseases that affect nutritional status

* Gastrointestinal diseases that affect the absorption of nutrites
* Cancer
* Chronic kidney disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 800 volunteers in total, men and women from 37 locations in Spain distributed in 8 different areas (Nielsen Areas) covering the eastern, eastern, eastern, southern, southern, central, northwestern, northern and metropolitan areas of Madrid and Barcelona in Spain.
  These 800 participants will be randomized according to sex and the territory to which they belong, into three age groups: one group will be between 60 and 70 years old, another group will be between 71 and 80 years old, and the third will be made up of people over 80 years old. In addition, 100 of these subjects must be regular consumers of omega-3 supplements.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
omega-3 index | At the time of enrollement
  The omega-3 index measure the presence of omega-3 fatty acids in the erythrocyte membrane

SECONDARY OUTCOMES:
Nutritional assesment | At the time of enrollement
  Food frecuency questionarie
Physical activity assesment | At the time of enrollement
  Physical activity questionaries
Socioeconomic assesment | At the time of enrollement
  Socioeconomic questionaries
DNA genotyping | At the time of enrollement
  Specific genes related to lipid metabolism and cardiovascular risk will be genotiped only in the validation cohort
Plasma triacylglycerides | At the time of enrollement
  Plasma triacylglycerides only in the validation cohort
Plasma cholesterol | At the time of enrollement
  Plasma Total cholesterol, HDL-Cholesterol, LDL-cholesterol only in the validation cohort
Plasma glucose | At the time of enrollement
  Plasma glucose levels only in the validation cohort
Plasma insulin | At the time of enrollement
  Plasma insulin levels only in the validation cohort

CONTACTS AND LOCATIONS:
Overall Officials: Estefanía Sánchez Rodríguez, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Avd del Conocimiento 19, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
all collected anonimous IPD
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: A proposal that describes planned analyses must be submitted, and a data sharing agreement must be signed. Researcher will contact the IP of tthe present project (estefaniasr@ugr.es), explain the proposal. She will send them an agreement document to be submitted.